CLINICAL TRIAL: NCT02418169
Title: Association Between Craniofacial Fractures and Brain Injuries: Diagnostic and Therapeutic Considerations
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: T74/2015
Record Dates: First submitted 2015-04-13; First posted 2015-04-16 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Brain Injuries; Skull Fractures
MeSH Terms: conditions — Brain Injuries; Skull Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- retrospective, severe traumatic brain injury: All patients in 2010-2014 with severe traumatic brain injury admitted to Turku University Central Hospital (TUCH)
- retrospective, craniofacial fracture: All patients in 2010-2014 with craniofacial fracture admitted to TUCH.
- prospective, severe traumatic brain injury: All patients in 2015-2017 with severe traumatic brain injury admitted to Turku University Central Hospital (TUCH)
- prospective, craniofacial fracture: All patients in 2015-2017 with craniofacial fracture admitted to TUCH.

SUMMARY:
This study evaluates the association between traumatic brain injuries and craniofacial or/and skull fractures. Purpose is to find out the amount of missed diagnoses and improve primary diagnostics of trauma patients.

DETAILED DESCRIPTION:
A part of mild TBIs remains undiagnosed. Therefore the primary diagnostics of trauma patients needs to be improved. According to some studies, a part of trauma patients' concomitant injuries weren't diagnosed in the emergency room (ER) but were diagnosed later in the clinics. In addition to difficult diagnostics the treatment of these patients demands close co- operation between many specialities.

The aim of this study is to evaluate the association between TBIs and facial fractures. The real amount of facial fractures in patients with severe TBI and the clinical significance of these fractures are evaluated. Also the number of patients with facial fractures and a concomitant TBI is evaluated. The aim is to find out the amount of patients with missed diagnoses. Other aims of are to determine the effect of the type or location of a facial fracture on the in- cidence and severity of TBI. With the help of the results it would be possible to improve the comprehensive diagnostics and early treatment of patients with a facial fracture or a TBI.

The retrospective and prospective data on patients with TBI and/or facial fracture are collect- ed at Turku University Hospital. The comparison of the two groups will give information on the amount of patients with missed diagnosis of TBI or facial fracture. The results can be utilised in planning strategy for comprehensive diagnostics and treatment of the patients. In the research group the investigators have specialists in the fields of oral and maxillofacial surgery, neurol- ogy and otorhinolaryngology.

ELIGIBILITY:
Inclusion Criteria:

* Severe traumatic brain injury, GCS 8 or less and/or Craniofacial fracture

Exclusion Criteria:

* Died before admitted to hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with severe traumatic brain injury, patients with craniofacial fractures
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
survival | 12 months